CLINICAL TRIAL: NCT03303326
Title: Arab American Women's Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Distinguished Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 064917B3E
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Mental Health Wellness 1
Keywords: sexual health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Interview (Experimental): A 60-minute interview about women's health conducted immediately after baseline questionnaires.
  Interventions: Behavioral: Immediate interview
- Delayed Interview (No Intervention): The interview is conducted after the follow-up questionnaires are completed, rather than after baseline.

INTERVENTIONS:
Behavioral: Immediate interview — A women's health interview that obtains information about physical, mental, and sexual health, particularly relatively private sexual health-related attitudes and experiences, as well as conflicts and stress related to sexuality.
  Other Names: Women's Health Interview
  Arms: Immediate Interview

SUMMARY:
This study evaluates how Arab American women's cultural values and sexual health are related to their physical and emotional health. The study will also examine whether engaging in a sexual health interview affects women's physical and emotional health.

DETAILED DESCRIPTION:
Sexuality is an important aspect of health, in part because emotional conflicts over sexuality as well as unwanted sexual experiences can impact physical and psychological health; yet no studies have examined sexual health among Arab American women in the U.S. These women face the task of negotiating their heritage culture and the American culture in which they reside. This may result in bicultural identity conflict for some women as they try to negotiate these two identities, which may have implications for sexuality and sexual health due to the two cultures' disparate views on sexuality. Confidential discussion of these sensitive topics with a knowledgeable interviewer may yield beneficial effects.

The overall goal of the current study is to fill the gap in the literature on Arab American sexual health by examining how sexual health is related to physical and psychological health. This will be accomplished using both: a) correlational findings about sexual, physical, and psychological health from information gathered through self-report questionnaires and a 60-minute women's health interview; and b) an experimental test of the effects of the women's health interview on physical and psychological health. A sample of young adult Arab American women will be assessed at baseline via questionnaires for various constructs (sexual attitudes, cultural and religious identity, and physical and mental health), and then randomized to either an immediate or delayed health interview, with a 5-week follow-up reassessment.

It is hypothesized that lower sexual well-being, negative sexual self-schemas, and unwanted sexual experiences will correlate with more somatic and psychological health symptoms and lower satisfaction with life. It is also hypothesized that participants who have the immediate interview will report greater reduction in somatic and psychological symptoms and a greater willingness to discuss sexual health with medical providers compared to participants who are not interviewed (i.e., have a delayed interview after follow-up assessment).

ELIGIBILITY:
Inclusion Criteria:

* Arab American or Chaldean
* Female
* Age 18-35

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire | Change from baseline to 5-week follow-up
  Physical symptoms

SECONDARY OUTCOMES:
Brief Symptom Inventory | Change from baseline to 5-week follow-up
  Psychological symptoms
Satisfaction with Life Scale | Change from baseline to 5-week follow-up
  Satisfaction with life
Sexual Self-Schema Scale | Change from baseline to 5-week follow-up
  Sexual self-schemas
Sexual Self Disclosure Scale (Catania) | Change from baseline to 5-week follow-up
  Self-reported ease or difficulty with disclosing information about sexuality
Sexual Self Disclosure Scale (Herold & Way) | Change from baseline to 5-week follow-up
  Degree of past sexual disclosure
Female Sexual Function Index | Change from baseline to 5-week follow-up
  Female sexual function
Sexual Satisfaction Scale for Women | Change from baseline to 5-week follow-up
  Sexual satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lumley, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No